CLINICAL TRIAL: NCT03261297
Title: Epidemiology of Chronic Diarrhea Among Children Admitted to Gastroenterology Unit at Assuit University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, moustafa abd ellatif, director clinical research, Assiut University
Other Study IDs: 17100287
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Chronic Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic diarrhea is defined as stool volume of more than 10g/kg/day in toddlers/infants and greater than 200 g/day in older children that lasts for 14 days or more.

Chronic diarrhea has many of causes can calcified as infectious & noninfectious causes.

* Infectious causes as: - Escherichia coli, Giardia Lamblia, tuberculosis, Clostridium difficile & Shigella.
* Noninfectious causes as(Abnormal digestive processes- Nutrient Mal -absorption- Immune/ inflammatory- Defects of electrolyte And metaboliteTransport- Motility disorders- Diarrhea associated With exogenous substances)

There are four basic pathophysiological categories of diarrhea: as ( osmotic diarrhea- secretory diarrheas- motility related diarrhea- Inflammatory diarrhea)

DETAILED DESCRIPTION:
Infectious diarrhea caused by invasive bacteria (Shigella, Salmonella, Campylobacter) or a cytotoxic organism result ting in mucosal histologic damage and inflammation (Entamoeba histolytica). (Hedberg etal., 1994)

Giardia lamblia Transmission is via the faecal oral route or via ingestion of contaminated water sources. Symptoms of Giardia infection include diarrhea, malaise, flatulence, foul smelling greasy stools, bloating/ distention and, less commonly, nausea, anorexia and vomiting. (Dib etal., 2008)

Entamoeba histolytica is the causative agent of amoebiasis. The majority of patients will have asymptomatic or low level disease with a gradual onset of diarrhea with generalized abdominal tenderness. Fever is not usually associated with amoebic disease. Mucus and/or blood may be present if the organism penetrates the bowel wall and causes mucosal damage. (Van Hal etal., 2007)

Inflammatory bowel diseases, including Crohn disease & ulcerative colitis ,cause chronic diarrhea that is often associated with abdominal pain, elevated inflammatory markers, and increased concentrations of fecal calprotectin. The severity of the symptoms is highly variable with a pattern characterized by long periods of well-being followed by exacerbations (Bunn etal., 2001)

Lactose is the sugar found in milk .Because lactose is not digested properly in the small intestine of individuals who are lactose intolerant; it passes whole into the large intestine or colon. Upon reaching the colon it is broken down by the normal colon bacteria. This breakdown results in the production of carbon dioxide and hydrogen gases. The gas production can lead to (Abdominal distension, excess gas and diarrhea, watery and explosive bowel movements, urgency). The severity of symptoms is usually proportional to the amount of the milk sugar ingested with more symptoms following a meal with higher milk sugar content. (Marsha, 2012).

There are four basic pathophysiological categories of diarrhea:

In osmotic diarrheas, osmotically active substances draw fluids from the plasma into the jejunum along the osmotic gradients through the highly permeable jejunal epithelium. Examples of chronic diarrhea due to an osmotic cause include malabsorption states such as celiac disease, bacterial overgrowth, osmotic laxatives including salts, and lactulose and maldigestion as occurs in disaccharidase deficiency and pancreatic exocrine insufficiency.Osmotic diarrheas might result in steatorrhea (passage of fat in to the stool). (Pardi etal., 2002)

In secretory diarrheas, there is secretion of isoosmolar fluid into the intestine. In this situation, other electrolyte abnormalities might coexist. Thus, hypokalemia and acidosis are associated with Verner-Morrison syndrome or VIPoma; Examples of secretory diarrheas include congenital abnormalities such as congenital chloridorrhea, in which an abnormality in the genetic control of chloride-bicarbonate exchange in the ileum results in the loss of chloride into the stool. (Long etal., 1981) Secretory diarrhea might be associated with altered motor functions induced by the hormone or transmitter produced by the tumor, as in carcinoid diarrhea. (Von etal., 1993) The typical features of secretory diarrhea include the persistence of the diarrhea with fasting and the absence of steatorrhea, hypokalemia and acidosis typically suggest VIPoma syndrome (Camilleri etal., 1982)

In motility related diarrhea, Motility disorders cause diarrhea by either accelerating gastrointestinal transit (e.g., post vagotomy diarrhea) or by slowing transit, thereby predisposing to small intestinal bacterial overgrowth (SIBO) (e.g., scleroderma).The most prevalent forms of motility-related diarrheas is IBS-D, Rapid small-bowel transit is a relatively common finding in patients with diabetes or autonomic neuropathies, or patients who have undergone upper gastrointestinal tract surgery. (Posserud etal., 2007)

In Inflammatory diarrhea occurs when there is damage to the mucosal lining or brush border, which leads to a passive loss of protein-rich fluids and a decreased ability to absorb these lost fluids. It can be caused by bacterial infections, viral infections, parasitic infections, or autoimmune problems. It can also be caused by tuberculosis, colon cancer, and enteritis (Camilleri etal., 2014)

ELIGIBILITY:
Inclusion Criteria:

* 1. -all patient from 1 month up to 17 years (1month-17 year) admitted gastroenterology unit at Assuit University Children Hospital 2. Diarrhea 14 days or more ( ≥14 day)

Exclusion Criteria:

* 1. age less than 1 month (≤1 month) 2. diarrhea less than 14 days (≤14 day) 3. chronic diarrhea due to malignancy & chemotherapy

Ages: 1 Month to 17 Years | Sex: All
Age Groups: Child
Study Population: epidemiological study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2018-08-22 (Estimated)

PRIMARY OUTCOMES:
Identify the prevalence of chronic diarrhea at Gastroenterology unit at Assuit University Children Hospital | one year
  Not yet recruiting: Participants are not yet being recruited

SECONDARY OUTCOMES:
improve hospital to meet the most common couse of diarrha in our hospital | one year
  Not yet recruiting: Participants are not yet being recruited

CONTACTS AND LOCATIONS:
Locations (1):
- Moustafa Abd Ellatif, Asyut, Egypt